CLINICAL TRIAL: NCT06334458
Title: Development of a New Algorithm to Integrate Clinical, Omics, DNA Methylation Biomarkers and Epidemiological Data for Early Detection of Pancreatic Cancer in High-risk Individuals
Brief Title: Epigenomic and Machine Learning Models to Predict Pancreatic Cancer
Acronym: IMAGene
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 1910
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Early Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early diagnosis for Pancreatic Cancers in high-risk asymptomatic subject groups (Other): Early diagnosis for pancreatic cancer in first degree healthy/asymptomatic relatives of patients with exocrine pancreatic cancer (high-risk asymptomatic subject groups)
  Interventions: Diagnostic Test: Early diagnosis for Pancreatic Cancers in high-risk asymptomatic subject groups

INTERVENTIONS:
Diagnostic Test: Early diagnosis for Pancreatic Cancers in high-risk asymptomatic subject groups — Early diagnosis for Pancreatic Cancers in high-risk asymptomatic subject groups by developing and validating a comprehensive cancer risk prediction algorithm (CRPA) as a clinical support tool to calculate a personalized risk profile

SUMMARY:
The goal of the multicentric and interdisciplinary IMAGene project is to pursue early diagnosis for Pancreatic Cancers in high-risk asymptomatic subject groups, by developing and validating a comprehensive cancer risk prediction algorithm (CRPA) as a clinical support tool to calculate a personalized risk profile.

The study is a longitudinal, non-randomized exploratory clinical study. A total of 170 asymptomatic first-degree relatives of PC patients.

DETAILED DESCRIPTION:
The study is a longitudinal, non-randomized exploratory clinical study. A total of 170 asymptomatic first-degree relatives of PC patients.

The study population consists of 170 first (1st) degree healthy/asymptomatic relatives of patients with exocrine pancreatic cancer, where the patient satisfies one OR more of the following conditions:

* was diagnosed with pancreatobiliary cancer <50 years of age;
* was diagnosed with pancreatobiliary cancer >50 years of age AND personal history of any solid cancers.

The CRPA will be assessed in 170 first degree relatives of PC patients, in whom the development of pancreatic cysts will be assessed by WB-MRI at baseline and at one year.

ELIGIBILITY:
Inclusion Criteria:

* 1st degree healthy/asymptomatic relatives of patients with exocrine pancreatic cancer, where the patient satisfies one OR more of the following conditions:

  * was diagnosed with pancreatobiliary cancer <50 years of age;
  * was diagnosed with pancreatobiliary cancer >50 years of age AND personal history of any of the following cancers: Breast cancer, Ovarian, fallopian tube or primary peritoneal cancer, Melanoma, Colorectal cancer, Endometrial cancer, Prostate cancer, Oesophagogastric cancer, Urinary tract cancer, Small bowel cancer, Brain tumour, Sebaceous skin tumour;
  * was confirmed diagnosis of any of the following conditions in the family: Hereditary Breast and Ovarian Cancer, Peutz-Jeghers syndrome, hereditary pancreatitis, Lynch Syndrome, Familial Atypical Multiple Mole Melanoma Syndrome;
  * significant family history in first degree relatives for cancer (e.g. two or more cancers in one individual or the same cancer in more individuals;
  * a single 1st degree relative with pancreatic cancer;
  * being a patient alive after 5 years from diagnosis (cancer free or currently treated).
* Cancer free at the time of enrollment;

Exclusion Criteria:

* Individuals with comorbidities that adversely influence their ability to tolerate the screening procedures or the screen-detected findings, or tolerate treatment of an early- stage screen-detected cancer, or that limit their life expectancy.
* Subjects already diagnosed with cancer currently in treatment;
* Subjects who are already in the process of clinical assessment or included in a screening program for a suspected tumour.
* Contraindications for the Whole-Body Magnetic Resonance Imaging (WB-MRI) radiological exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Observation of a two or three-fold enrichment in early detection of suspicious pancreatic lesion using the CRPA algorithm | 5 years
  Develop/calibrate/validate a comprehensive cancer risk prediction algorithm (CRPA) and observe a two or three-fold enrichment in early detection of suspicious pancreatic lesion in our sample of HR individuals (incidence about 24%), stratified through the application of the Machine Learning algorithm, the CRPA.
Identification of one or more abnormal methylation changes present in blood cells of participants with suspicious lesions versus methylation profiles of participants with no identified lesions | 5 years
  Provide evidence that the implementation of epigenetic biomarkers profiles in CRPA leads to a significant improvement of accuracy of cancer risk prediction models.
  This endpoint will be reached with the identification of a methylation profile referred to as a risk signature (defined as one or more abnormal methylation changes present in blood cells of participants) by analyzing blood cells methylation profiling data from participants with suspicious lesions vs methylation profiles of participants with no identified lesions;
Validation of igenetic biomarker testing in liquid biopsy followed by radiological exam as early cancer diagnostic tool | 5 years
  Validate whether the use of epigenetic biomarker testing in liquid biopsy followed by radiological exam can be an early cancer diagnostic tools for PC in High Risk (HR) subjects

CONTACTS AND LOCATIONS:
Overall Officials: Serena Oliveri, Principal Investigator — European Institute of Oncology
Locations (4):
- Toulouse University Hospital, Toulouse, France
- European Institute of Oncology, Milan, Italy
- Oncological Institute "Prof. Dr. Ion Chiricuta", Cluj-Napoca, Romania
- Catalan Institute of Oncology, Barcelona, Spain